CLINICAL TRIAL: NCT03294252
Title: Phase I / II Dose Escalation of Oxaliplatin Via a Laparoscopic Approach of Aerosol Pressurized Intraperitoneal Chemotherapy for Nonresectable Peritoneal Metastases of Digestive Cancers (Stomach, Hail and Colorectal)
Brief Title: Oxaliplatin in PIPAC for Nonresectable Peritoneal Metastases of Digestive Cancers
Acronym: PIPOX
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The 34 patients included had all completed their treatment period under the protocol and the data could be collected to assess the main objective and the secondary objectives before the last theoretical follow-up.
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICO-N-2016-03
Record Dates: First submitted 2017-09-22; First posted 2017-09-27 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Digestive Cancer
Keywords: PIPAC; oxaliplatin; peritoneal metastases
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — Fluorouracil; Leucovorin; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oxaliplatin (Experimental): The experimental drugs used in this protocol are Oxaliplatin, 5-Fluorouracil and L-Folinic acid. All are used as part of their marketing authorization, with the exception of Oxaliplatin as regards its mode of administration specific to the PIPAC procedure (injection and nebulisation in intraperitoneal).
  Interventions: Drug: 5-Fluorouracil; Drug: L-Folinic acid; Drug: Oxaliplatin

INTERVENTIONS:
Drug: 5-Fluorouracil — Presentation: Concentrated solution for concentrated infusion in vials containing 250 mg, 500 mg, 1 g and 5 g, in 5 ml, 10 ml, 20 ml and 100 ml respectively, providing a 50 mg / ml solution. Dosage: 400mg / m2. Administration: IV. Day of administration: between 1 h and 24 h before PIPAC.
Drug: L-Folinic acid — Presentation: lyophilisate for parenteral use, dosed at 25 mg, and in the form of a solution for injection by IM or IV dosed at 25 mg / 2.5 ml. Dosage: 20mg / m2. Administration: IV. Day of administration: between 1 h and 24 h before PIPAC.
  Other Names: ELVORIN
Drug: Oxaliplatin — Concentrated solution for infusion dosed with 50 mg and 100 mg. Dosage: depending on the dose range assigned to inclusion (from 90mg / m2 to 300mg / m2). Administration: the solution is packaged in a syringe which is subsequently used for injection and not in a conventional bag. The product is administered in a high-pressure injector, during the PIPAC. Day of administration : J1 of PIPAC

SUMMARY:
Current curative treatment of digestive peritoneal carcinomatosis consists of complete cytoreduction surgery associated with intraperitoneal chemotherapy. This treatment has important limits: a high morbimortality and the impossibility of repeating the sessions. The majority of patients are therefore treated with systemic chemotherapy, which despite its progress, remains palliative.

Pressurized Intraperitoneal aerosol chemotherapy (PIPAC) has many advantages: under laparoscopy, low morbidity, good intratumoral penetration of cytotoxics, possibility of repeating the sessions and low financial cost.

Therefore, the investigator propose a phase 1 study, in colorectal and stomach cancer, with oxaliplatin doses escalation in Pressurized Intraperitoneal aerosol chemotherapy. It would allow a better tumor response, with potentially few risks and thus improve survival in patients with digestive peritoneal carcinoses, increasing access to cytoreductive surgery.

DETAILED DESCRIPTION:
The objective of this study is to determine the maximum tolerated dose (mtd) of oxaliplatin to be used during PIPAC.

Study design is a phase I/II, multicentre, non-comparative, non-randomised dose escalation clinical trial.

The phase I study will consist of a 3 by 3 dose escalation according to modified fibonacci dose escalation, starting at the current PIPAC dose (i.e. 90mg/m2), up to a maximum dose of 300mg/m2, corresponding to the current Intraperitoneal chemohyperthermia.

Each patient may receive up to 5 PIPAC sessions ; DLT period will be from the first day (D1) of the first PIPAC session until the end of the second PIPAC session, including the interval chemotherapy (i.e. D-1 of the 3rd CIPPA session), i.e. 4 to 6 weeks later ; Phase II study is an extension cohort at the recommended dose determined in the Phase I study. It will be a multi-centre, single-arm study and will analyse overall patient survival and secondary resectability rates with complete cytoreductive surgery and intraperitoneal chemohyperthermia. It will be conducted in approximately 20 patients treated at the recommended dose and followed for 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age ≥ 18 years 2. Histological or cytological diagnosis or suspicion of peritoneal carcinosis of colorectal, gastric or bowel origin 3. Having previously received at least 3 months of systemic chemotherapy for metastatic disease (type of chemotherapy left to the discretion of each investigator). Patients who received bevacizumab (Avastin®) can be included if and only if the time between the last treatment administered and the first PIPAC received is at least 4 weeks 4. ECOG performance index < or = 2 5. Life expectancy> 3 months 6. Peripheral neuropathy grade ≤ 1 7. Hematological function: Hemoglobin ≥ 9 g / dL, leukocytes ≥ 4000 / mm3, PNN ≥ 1500 / mm3, platelets ≥ 100 000 / mm3 8. Creatinine clearance> 50 mL / min (cockcroft and Gault formula) 9. Hepatic function: Total bilirubin ≤ 1.5 x ULN, ASAT and ALAT ≤ 3 x ULN, Alkaline phosphatases ≤ 3 x ULN 10 . Patients with no known or partial deficiency of Dihydropyrimidine dehydrogenase (i.e. DPD) 11. Effective contraception for women of childbearing age 13. Informing the patient and obtaining free, informed and written consent signed by the patient and his / her investigator.

14. Affiliated subject or beneficiary of the social security scheme.

Exclusion Criteria:

1. Patients who received bevacizumab (Avastin®) less than 4 weeks ago can not be included
2. Extra-peritoneal metastases, except for less than 3 pulmonary nodules (each size <5mm)
3. Known hypersensitivity to Oxaliplatin
4. Known complete dihydropyrimidine dehydrogenase (i.e. DPD) deficiency
5. Peripheral neuropathy Grade >1 due to or not with Oxaliplatin previously used
6. Active or other serious underlying disease that may prevent the patient from receiving treatment
7. Intracranial or intraocular hypertension (ongoing at the time of inclusion)
8. Severe or Severe Heart Failure (ongoing at the time of inclusion)
9. Complete intestinal obstruction (ongoing at the time of inclusion)
10. Other concurrent cancer or history of cancer other than in situ cancer of treated cervix or basal cell carcinoma or squamous cell carcinoma
11. Pregnant or nursing women
12. Persons deprived of their liberty or under guardianship or unable to give their consent
13. Inability to submit to medical follow-up of the trial for geographical, social or psychological reasons
14. Long-term corticosteroids (duration> 3 months), except for weaning for at least 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2019-02-05 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Maximal Tolerated Dose | 8 to 12 weeks
  Maximal tolerated dose 3x3 patients inclusion(modified fibonacci dose escalation)
Recommanded dose for the extension phase | 8 to 12 weeks
  Dose level below the maximum tolerated dose

SECONDARY OUTCOMES:
Cumulative toxicity after the end of the PIPAC sessions received (maximum 5) at the same dose level | 24 months after the last PIPAC received
  with CTC-AE scale
Overall survival | 24 months after the last PIPAC received
  Median overall survival at the end of the study
Progression-Free Survival | 12 months after the last PIPAC received
  Median PFS, time between the first PIPAC received and progression or death in absence of progression

CONTACTS AND LOCATIONS:
Overall Officials: DUMONT Frederic, MD, Principal Investigator — Institut de Cancérologie de l'Ouest
Locations (3):
- France (3):
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - ICO René Gauducheau, Saint-Herblain
  - Hopital Begin, Saint-Mandé

REFERENCES:
- [Derived] Dumont F, Passot C, Raoul JL, Kepenekian V, Lelievre B, Boisdron-Celle M, Hiret S, Senellart H, Pein F, Blanc-Lapierre A, Raimbourg J, Thibaudeau E, Glehen O; BIG-RENAPE Networks. A phase I dose-escalation study of oxaliplatin delivered via a laparoscopic approach using pressurised intraperitoneal aerosol chemotherapy for advanced peritoneal metastases of gastrointestinal tract cancers. Eur J Cancer. 2020 Nov;140:37-44. doi: 10.1016/j.ejca.2020.09.010. Epub 2020 Oct 8. PMID 33039812
- [Derived] Dumont F, Senellart H, Pein F, Campion L, Glehen O, Goere D, Pocard M, Thibaudeau E. Phase I/II study of oxaliplatin dose escalation via a laparoscopic approach using pressurized aerosol intraperitoneal chemotherapy (PIPOX trial) for nonresectable peritoneal metastases of digestive cancers (stomach, small bowel and colorectal): Rationale and design. Pleura Peritoneum. 2018 Sep 15;3(3):20180120. doi: 10.1515/pp-2018-0120. eCollection 2018 Sep 1. PMID 30911664